CLINICAL TRIAL: NCT05532410
Title: Optic Disc Photograph Collection Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT1085
Record Dates: First submitted 2022-09-02; First posted 2022-09-08 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Retina Disease; Glaucoma; Normal
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Fundus Camera (Other)
  Interventions: Device: Fundus Camera

INTERVENTIONS:
Device: Fundus Camera — The fundus camera is suitable for photographing, displaying and storing data relating to the retina and surrounding parts of the eye. These photographs assist with the diagnosis and follow-up of eye diseases, which can be visually monitored and photographically documented.

SUMMARY:
The objective of this study is to collect stereo-optic disc photographs for potential future analysis.

ELIGIBILITY:
Inclusion Criteria

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects met inclusion/exclusion criteria for the OPT1060 protocol

Exclusion Criteria

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects not able to obtain acceptable OCT, Stereo, or Optomap images due to ocular media opacity or other reasons

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Bland-Altman Plots of Stereo Disc Photos, SLO images and OCT Scans | 1 year
Deming Regression of Stereo Disc Photos, SLO images and OCT Scans | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois College of Optometry, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No